CLINICAL TRIAL: NCT01439711
Title: Phase II Study of Neoadjuvant Letrozole for Postmenopausal Women With Estrogen Receptor Positive Ductal Carcinoma In SITU (DCIS)
Brief Title: Letrozole in Treating Postmenopausal Women With Ductal Carcinoma in Situ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-40903; CDR0000701992 (Registry Identifier: Physician Data Query); U10CA037447 (NIH); NCI-2011-03452 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; estrogen receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- letrozole + MRI + surgery (Experimental): Patients receive letrozole (2.5 mg) one tablet each day after confirmation that the MRI is acceptable. There is a 3 and 6 month disease evaluation by MRI of both breasts. If the DCIS has grown, the patient will have surgery to remove it and will continue to take letrozole until the day before surgery. It is expected that decisions regarding any adjuvant treatment will be made individually based on best practice guidelines, using informed and shared decision making between the patient and provider.
  Interventions: Drug: letrozole; Procedure: MRI; Procedure: conventional surgery

INTERVENTIONS:
Drug: letrozole
Procedure: MRI
Procedure: conventional surgery

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by blocking the use of estrogen by the tumor cells or by lowering the amount of estrogen the body makes.

PURPOSE: This phase II trial is studying how well letrozole works in treating women with ductal carcinoma in situ.

DETAILED DESCRIPTION:
Treatment with letrozole begins within 21 days of registration, and only after notification has been received from the UCSF Breast MRI Research Laboratory that the baseline MRI is acceptable. Protocol therapy will consist of 6 months of letrozole, administered orally at a dose of 2.5 mg/day. Patients will have a MRI for disease evaluation at months 3 and 6. All patients will continue to take study drug until the day prior to surgery, whether at month 3 or at month 6 or may stop if they experience unacceptable toxicity. It is expected that decisions regarding any adjuvant treatment (eg, radiation and hormonal therapy) will be made individually based on the best practice guidelines, using informed and shared decision making between patient and provider. The primary and secondary objectives are provided below.

Primary objective:

1. To estimate the mean change in MRI tumor volume from pretreatment to completion of preoperative endocrine therapy in estrogen receptor-positive (ER+) ductal carcinoma in situ (DCIS), as well as to determine whether 3-month change in volume correlates with 6-month change.

Secondary objectives:

1. To assess radiographic-pathologic correlation between MRI findings and histopathology, including the prevalence of occult invasive cancer in patients undergoing neoadjuvant endocrine therapy for DCIS.
2. To compare changes in MRI maximum lesion diameter and mammographic extent at baseline and following treatment. These are two additional radiographic parameters which may also biological response to therapy.
3. To determine practice patterns of adjuvant hormonal and radiation therapy in patients who complete neoadjuvant letrozole therapy for DCIS.
4. To determine whether Ki67 is reduced with neoadjuvant letrozole treatment for DCIS, and to compare the reduction in proliferation between radiographic responders and non-responders.
5. To identify baseline IHC and expression biomarkers predictive of response to treatment, with response determined by extent of Ki67 reduction. Subsets showing the greatest reduction in Ki67 would be the most likely candidates for non-operative treatment in future studies.
6. To examine whether germline polymorphisms are associated with clinical endpoints, including treatment-related toxicity or efficacy outcomes, or with expression of biomarkers in serum or tumor.
7. To assess quality-of-life and musculoskeletal symptoms associated with neoadjuvant letrozole for ER positive DCIS.

Patients will be followed up to 6 months post-surgery.

ELIGIBILITY:
Eligibility Criteria:

1. Histologic documentation: Pathologic confirmation of ductal carcinoma in situ (DCIS) of the female breast without invasive cancer, with diagnosis rendered on core biopsy only, completed within 60 days before registration. Patients diagnosed with DCIS on the basis of surgical biopsy are not eligible for this study.

   1. Patients with microinvasion on diagnostic core biopsy, defined as tumor ≤ 1 mm in greatest dimension, will be allowed to participate.
   2. All patients must have a clip placed, either at the time of the diagnostic biopsy or at the time of the baseline MRI prior to the start of treatment.
2. Tissue samples: Patient has diagnostic tissue available for correlative studies.
3. Clinical stage: Tis or T1mi N0, M0
4. Hormone receptor status: DCIS must express estrogen and/or progesterone receptor, as determined by immunohistochemical methods on the diagnostic pathology sample, according to the local institution's standard protocol. Greater than or equal to 1% cells will be considered to be positive.
5. Menopausal status: Patients must be postmenopausal defined as:

   1. Age ≥ 55 years and one year or more of amenorrhea
   2. Age < 55 years and one year or more amenorrhea, with an estradiol assay < 20pg/ml
   3. Surgical menopause with bilateral oophorectomy (at least 28 days must elapse from surgery to time of study registration)

   The use of GnRH analogs to achieve post menopausal status is not allowed.
6. Prior treatment:

   1. No prior surgical excision in the index breast for current DCIS diagnosis of DCIS
   2. Any exogenous hormone therapy must be completed 4 weeks prior to registration
   3. Any patients with a history of tamoxifen or raloxifene use within two years of current DCIS diagnosis are not eligible
   4. No prior neoadjuvant/adjuvant therapy for current DCIS diagnosis
7. Contraindication to MRI: No contraindications to breast MRI
8. Measurable disease: Mammographic extent of calcifications must be accurately measurable in at least one dimension with each lesion ≥ 1 cm and ≤ 7 cm

   1. DCIS must be visible on MRI based on central review.
   2. Patients with palpable DCIS or adenopathy are not eligible to participate.
   3. Patients with multifocal or bilateral disease are eligible.
9. History of osteoporosis: Women diagnosed with osteoporosis may participate in this trial provided they are receiving appropriate therapy or if they have declined therapy.
10. Age: Patients ≥ 18 years of age
11. Performance Status: ECOG performance status 0 or 1
12. Pregnancy/nursing status: Not pregnant or nursing
13. Required Initial Laboratory Values:

    1. ANC ≥ 1,000/μL
    2. Platelet count ≥ 100,000/μL
    3. Serum creatinine ≤ 1.7 mg/dL
    4. Bilirubin ≤ 2.0 mg/dL
    5. AST/ALT ≤ 2.5 times upper limit of normal
    6. Serum estradiol level assay < 20 pg/mL *Required for patients < 55 years of age and one year or more of amenorrhea

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Hwang, MD, MPH, Study Chair — Duke University
Locations (32):
- United States (32):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Bay Area Tumor Institute, Oakland, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Saint Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Northwest Hospital Center, Randallstown, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Sparrow Hospital, Lansing, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - M. D. Anderson Cancer Center, Houston, Texas
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Hospitals, Norfolk, Virginia

REFERENCES:
- [Derived] Marks JR, Zhang D, Hardman T, Chen YY, Hall A, Simpson L, Hieken T, Bedrosian I, Price E, Sheng J, Dai Y, Lee M, Sibley AB, Owzar K, Hwang ES. Genomic alterations are associated with response to aromatase inhibitor therapy for ER-positive postmenopausal ductal carcinoma in situ: (CALGB 40903, Alliance). Breast Cancer Res. 2025 Feb 20;27(1):26. doi: 10.1186/s13058-025-01963-5. PMID 39980051
- [Derived] Hwang ES, Hyslop T, Hendrix LH, Duong S, Bedrosian I, Price E, Caudle A, Hieken T, Guenther J, Hudis CA, Winer E, Lyss AP, Dickson-Witmer D, Hoefer R, Ollila DW, Hardman T, Marks J, Chen YY, Krings G, Esserman L, Hylton N. Phase II Single-Arm Study of Preoperative Letrozole for Estrogen Receptor-Positive Postmenopausal Ductal Carcinoma In Situ: CALGB 40903 (Alliance). J Clin Oncol. 2020 Apr 20;38(12):1284-1292. doi: 10.1200/JCO.19.00510. Epub 2020 Mar 3. PMID 32125937

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole + MRI: Protocol Therapy will consist of 6 months of letrozole, administered orally at a dose of 2.5 mg/day. Patients will have a bilateral MRI for disease evaluation at months 3 and 6.
Period: Overall Study
Arm/Group | Letrozole + MRI
Started | 108
Completed | 68
Not Completed | 40
Not completed — Ineligible | 13
Not completed — Cancel | 3
Not completed — Progression Prior to Beginning Tx | 1
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 3
Not completed — Progression During Active Tx | 3
Not completed — Noncompliance | 3
Not completed — No MRI | 9

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Total MRI Functional Tumor Volume (FTV) Change From Baseline to Month 3 (V3)
Description: Mean total MRI FTV change from baseline to month 3 (V3): For patients with more than one measureable lesion on the MRI, the sum over all measureable lesions on the MRI was calculated at each time point. V3 was calculated by subtracting the total MRI FTV measured (i.e. the sum over all lesions present with MRI FTV measurements) at 3 months from the total MRI FTV measured at baseline. For V3 the raw change in the volume will be calculated for each patient and a mean and 95% confidence interval will be constructed using two-sided t-tests.
Time Frame: up to 3 months from start of treatment
Measure: Mean (95% Confidence Interval); unit: cubic centimeters
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 68
cubic centimeters | -1.93 [-2.87 to -0.98]
Statistical Analysis 1: Comparison: Letrozole + MRI; Test type: Superiority; p < 0.001, t-test, 2 sided

2. Primary Outcome: Mean Total MRI Functional Tumor Volume (FTV) Change From Baseline to Month 6 (V6)
Description: Mean total MRI FTV change from baseline to month 6 (V6): For patients with more than one measureable lesion on the MRI, the sum over all measureable lesions on the MRI was calculated at each time point. V6 was calculated by subtracting the total MRI FTV measured at 6 months from the total MRI FTV measured at baseline. For V6 the raw change in the volume will be calculated for each patient and a mean and 95% confidence interval will be constructed using two-sided t-tests.
Time Frame: up to 6 months from start of treatment
Measure: Mean (95% Confidence Interval); unit: cubic centimeters
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 68
cubic centimeters | -1.82 [-2.75 to -0.9]
Statistical Analysis 1: Comparison: Letrozole + MRI; Test type: Superiority; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Mean Total MRI Tumor Diameter Change From Baseline to Month 3
Description: To ascertain the change in maximum tumor diameter from baseline to 3 months (D3) the same methods as in Primary outcome #1 will be used but on diameter instead of volume. For patients with more than one lesion longest diameter measurement, the sum of all lesion longest diameter measurements was calculated.
Time Frame: 3-months
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 68
millimeters | -10.3 [-13.94 to -6.66]

4. Secondary Outcome: Change in Maximum Diameter at 6-months Based on Mammographic Measurement (MD6)
Description: Change in maximum diameter at 6-months based on mammographic measurement (MD6) will be estimated using the methods in Primary Outcome #1, but using the mammographic measurements instead.
Time Frame: 6-months
Population: Patients who completed a mammogram at both time points (baseline and month 6) with measurements available were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 52
millimeters | -3.31 [-7.0 to 0.38]

5. Secondary Outcome: Type of Primary Surgery (Mastectomy or Lumpectomy)
Description: Rate of Mastectomy will be estimated as the number of mastectomies divided by the number of surgeries. A 95% confidence interval will be constructed using exact binomial methods. Rate of Lumpectomy will be estimated as the number of lumpectomies divided by the number of surgeries. A 95% confidence interval will be constructed using exact binomial methods.
Time Frame: up to 6 months
Population: Patients who underwent surgery were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of surgeries
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 59
percentage of surgeries
  Rate of Mastectomy | 7 [2 to 16]
  Rate of Lumpectomy | 93 [84 to 98]

6. Secondary Outcome: Number of Re-excisions Required to Obtain Clear Margins
Time Frame: 3-months and 6-months
Reporting Status: Not Posted

7. Secondary Outcome: Extent of Residual DCIS Post Surgery
Time Frame: Up to 6 months post-surgery
Reporting Status: Not Posted

8. Secondary Outcome: Presence of Invasive Cancer at Surgery
Time Frame: 3-months and 6-months
Reporting Status: Not Posted

9. Secondary Outcome: Size of Margins (Smallest) at Surgery
Time Frame: 3-months and 6-months
Reporting Status: Not Posted

10. Secondary Outcome: Incidence of Toxicity as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. The percentage of patients with a maximum grade 3 or higher adverse event at least possibly related to the study treatment are reported below.
Time Frame: Up to 6 months post surgery
Population: Patients who had completed the study and had an Adverse Event Form submitted were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 67
Participants
  Allergic reaction | 31
  Cholesterol high | 7
  Gastrointestinal disorder | 2
  Hot flashes | 1

11. Secondary Outcome: Mean Total MRI Tumor Diameter Change From Baseline to Month 6
Description: Mean total MRI tumor diameter change from baseline to month 6: To ascertain the change in maximum tumor diameter from baseline to 6 months (D6) the same methods as in Primary Outcome #2 will be used but on diameter instead of volume.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 68
millimeters | -16.66 [-21.09 to -12.23]

12. Secondary Outcome: Mean Total MRI Tumor Diameter Change From Baseline to Month 6
Description: To ascertain the change in maximum tumor diameter from baseline to 6 months (D6) the same methods as in Primary outcome #2 will be used but on diameter instead of volume. For patients with more than one lesion longest diameter measurement, the sum of all lesion longest diameter measurements was calculated.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Letrozole + MRI
Number analyzed (Participants) | 68
millimeters | -16.66 [-21.09 to -12.23]

ADVERSE EVENTS:
Arm/Group | Letrozole + MRI
Serious Adverse Events (participants affected / at risk) | 2/90
Other Adverse Events (participants affected / at risk) | 75/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole + MRI (N=90)
Heart failure (Cardiac disorders) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole + MRI (N=90)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 3 (5)
Fracture (Injury, poisoning and procedural complications) | 3 (3)
Cholesterol high (Investigations) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 (87)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (28)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 (8)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hot flashes (Vascular disorders) | 50 (103)
Hypertension (Vascular disorders) | 16 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes